CLINICAL TRIAL: NCT04190550
Title: A Phase 1b Study With Expansion Cohort of Escalating Doses of KRT-232 (AMG 232) Administered in Combination With Standard Induction Chemotherapy (Cytarabine and Idarubicin) in Newly Diagnosed Acute Myelogenous Leukemia (AML)
Brief Title: Testing the Addition of an Anti-cancer Drug, Navtemadlin, to the Usual Treatments (Cytarabine and Idarubicin) in Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-08137; NCI-2019-08137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-115; 10367 (Other: City of Hope Comprehensive Cancer Center LAO); 10367 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; 4-demethoxydaunorubicin bis(hydrazone); navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (navtemadlin, cytarabine, idarubicin) (Experimental): Patients receive navtemadlin PO QD on days 1-7, cytarabine IV BID over 3 hours on days 1-7, and idarubicin IV over 10-15 minutes on days 1-3. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with residual disease may receive cytarabine IV BID over 3 hours for 5 days and idarubicin IV over 10-15 minutes for 2 days starting between days 14-21 of cycle 1 or the second cycle of navtemadlin, cytarabine, and idarubicin. Patients who achieve a CR or a CRi in either cycle 1 or 2 may receive cytarabine IV BID over 3 hours on days 1, 3, and 5 for 3-4 additional 28 to 35-day cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Idarubicin Hydrochloride; Drug: Navtemadlin

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Idarubicin Hydrochloride — Given IV
  Other Names: Idamycin; Idamycin PFS; Idarubicin HCl; IMI-30; SC-33428; Zavedos
Drug: Navtemadlin — Given PO
  Other Names: (3R,5R,6S)-5-(3-Chlorophenyl)-6-(4-chlorophenyl)-3-methyl-1-((1S)-2-methyl-1-(((1-methylethyl)sulfonyl)methyl)propyl)-2-oxo-3-piperidineacetic Acid; AMG 232; AMG-232; KRT 232; KRT-232; KRT232; MDM2 Inhibitor KRT-232

SUMMARY:
This phase Ib trial studies the side effects and best dose of navtemadlin when given together with the standard chemotherapy drugs cytarabine and idarubicin in patients with acute myeloid leukemia. Navtemadlin may stop the growth of cancer cells by blocking a protein called MDM2 that is needed for cell growth. Chemotherapy drugs, such as cytarabine and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving navtemadlin with cytarabine and idarubicin may stabilize cancer for longer when compared to giving usual treatments alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the toxicities of navtemadlin (KRT-232 [AMG 232]), cytarabine and idarubicin hydrochloride (idarubicin), and to determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of KRT-232 (AMG 232), cytarabine and idarubicin.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the pharmacokinetic (PK) profiles of KRT-232 (AMG 232), cytarabine and idarubicin when used in combination.

III. To evaluate p53 signaling induced by KRT-232 (AMG 232), cytarabine and idarubicin.

IV. To correlate KRT-232 (AMG 232), cytarabine and idarubicin exposure with pharmacodynamics endpoints (efficacy, toxicity, changes in p53 signaling).

EXPLORATORY OBJECTIVES:

I. To evaluate the response rate (RR) and progression free survival (PFS) of KRT-232 (AMG 232), cytarabine and idarubicin in acute myeloid leukemia (AML).

II. To evaluate potential predictive biomarkers, including MTF2 and H3K27me3, of response to KRT-232 (AMG 232), cytarabine and idarubicin in AML.

III. To evaluate the pharmacodynamic (PD) effects of KRT-232 and induction chemotherapy in AML blasts.

OUTLINE: This is a dose-escalation study of navtemadlin.

Patients receive navtemadlin orally (PO) once daily (QD) on days 1-7, cytarabine intravenously (IV) twice daily (BID) over 3 hours on days 1-7, and idarubicin IV over 10-15 minutes on days 1-3. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with residual disease may receive cytarabine IV BID over 3 hours for 5 days and idarubicin IV over 10-15 minutes for 2 days starting between days 14-21 of cycle 1 or the second cycle of navtemadlin, cytarabine, and idarubicin. Patients who achieve a complete response (CR) or a CR with incomplete hematologic recovery (CRi) in either cycle 1 or 2 may receive cytarabine IV BID over 3 hours on days 1, 3, and 5 for 3-4 additional 28 to 35-day cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and previously untreated AML (except acute promyelocytic leukemia [APL]) (>= 20% blasts in bone marrow or extramedullary leukemia) according to the World Health Organization (WHO), 2016 criteria. Note that patients who have received treatment with hypomethylating agents alone or in combination with venetoclax, ivosidenib or enasidenib for myelodysplastic syndrome (MDS) and have now transformed to AML are eligible.
* Eligible patients must show evidence of wild-type (WT) p53 as assessed by deoxyribonucleic acid (DNA) sequencing before initiation of KRT-232 (AMG 232).
* Patients must be considered candidates for intensive chemotherapy treatment with standard doses of cytarabine and idarubicin ("7+3 regimen").
* Left ventricular ejection fraction (LVEF) >= 50% as assessed by echocardiogram or radionuclide angiography.
* All non-hematological adverse events of any prior chemotherapy, surgery, or radiotherapy, except alopecia, must have resolved to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade =< 2 prior to starting therapy.
* Patient must be willing to submit the blood sampling and bone marrow sampling for the PK and PD analyses and exploratory biomarkers.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%).
* Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN), OR international normalized ratio (INR) < 1.5.
* Total bilirubin =< 2 mg/dl, unless from hemolysis, Gilbert's syndrome or liver infiltration with leukemia.
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN (=< 5 x ULN if liver infiltration with leukemia).
* Alkaline phosphatase (ALP) < 2.0 x ULN (if liver or bone metastases are present, < 3.0 x ULN)
* Creatinine within reference laboratory ranges OR glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 (by the Cockcroft Gault equation), with normalization to the patient's body surface area.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients with known leukemic involvement of the central nervous system (CNS) are eligible if, in the opinion of the treating physician, they are eligible for induction chemotherapy. These patients can receive the intrathecal treatment concurrently with the study treatment on protocol.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of KRT-232 (AMG 232) on the developing human fetus are unknown. For this reason and because MDM2 inhibiting agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation through 5 weeks (women) after receiving the last dose of KRT-232 (AMG 232). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of KRT-232 (AMG 232) administration. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug. Adequate methods of effective birth control include sexual abstinence (men, women); vasectomy; or a condom with spermicide (men) in combination with barrier methods, hormonal birth control or intrauterine device (IUD) (women).
* Female patients with child-bearing potential must have a negative serum pregnancy test within 72 hours prior to the first study drug administration.
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible.

Exclusion Criteria:

* Patients with evidence of p53 mutation or deletion (e.g. chromosome 17p deletion).
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 2) with the exception of alopecia.
* Patients receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy within 14 days of first receipt of study drug with the exception of: Hydroxyurea (HU) in patients who need to continue this agent to maintain white blood cell (WBC) count =< 50,000/mm^3.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to KRT-232 (AMG 232) or other agents used in study.
* Patients with uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia; patients receiving an anti-microbial agent may be eligible if the patient remains hemodynamically stable for 72 hours; patients with myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association [NYHA] class III and higher), unstable angina, or cardiac arrhythmia requiring medication are excluded.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because KRT-232 (AMG 232) is an MDM2 inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with KRT-232 (AMG 232), breastfeeding should be discontinued if the mother is treated with KRT-232 (AMG 232). These potential risks may also apply to other agents used in this study.
* Patients with reproductive potential not willing to use effective methods of contraception.
* Patients with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
* Patients with history of bleeding diathesis.
* Positive hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B), positive hepatitis total core antibody with negative HBsAG (suggestive of occult hepatitis B), or detectable hepatitis C virus ribonucleic acid (RNA) by a polymerase-chain reaction (PCR) assay (indicative of active hepatitis C - screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive).
* All herbal medicines (e.g., St. John's wort), vitamins, and supplements consumed by the subject within the 30 days prior to receiving the first dose of AMG 232, and continuing use, if applicable, will be reviewed by the principal investigator. Patients may continue to take all herbal medicines (e.g., St. John's wort), vitamins, and supplements if approved by the principal investigator.
* Use of any known CYP3A4 substrates with narrow therapeutic window (such as alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, sirolimus, or terfanide) within the 14 days prior to receiving the first dose of AMG 232 is not permitted. Other medications (such as fentanyl and oxycodone) may be allowed per investigator's assessment/evaluation. Use of any known CYP2C8 substrates with a narrow therapeutic window within the 14 days prior to receiving the first dose of KRT-232 (AMG 232) is not permitted.
* Use of any medications considered inhibitors or substrates of UGT1A1, or inhibitors or inducers of P-glycoprotein (gp) are not permitted. Caution should be used with concomitant antacids or proton pump inhibitor (PPI) products.
* Major surgery within 28 days of study day 1.
* Current use of warfarin, factor Xa inhibitors and direct thrombin inhibitors. Note: Low molecular weight heparin and prophylactic low dose warfarin are permitted. PT/PTT must meet the inclusion criteria. Subjects taking warfarin must have their INR followed closely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last dose of navtemadlin
  Toxicity will be coded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Based on the toxicity observed, a derived variable, the occurrence of dose limiting toxicity, will be created. Toxicities will be tabulated and reported according to dose level, grade, type, cycle, and attribution and, if numbers permit, by whether the patient had newly diagnosed or previously treated acute myeloid leukemia (AML). Cumulative incidence curves will be used to estimate the proportion of patients who will discontinue therapy for reasons of toxicity or general inability to tolerate the regimen. The data from all patients treated at the recommended phase 2 dose (RP2D), will be combined for a final summary and listing of toxicities observed.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of navtemadlin in combination with cytarabine and idarubicin | Pre-treatment and 1, 3, 5, 8, and 24 hours post-treatment on cycle 1, day 1 (1 cycle = 28-35 days)
  Will be quantitatively measured using liquid chromatography/tandem mass spectrometric (LC/MS/MS) method developed by the Analytical Pharmacology Core Laboratory at the Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins. For navtemadlin, the individual PK parameters from a single dose will be estimated for concentration maximum (Cmax), area under the curve (AUC), half-life (T1/2), apparent clearance (Cl/F), and apparent volume of distribution (V/F) using non-compartmental or compartmental PK methods with the software WinNonlin. Advanced population PK methods may be employed to assess the link between drug exposure and biological effects and efficacy.

OTHER OUTCOMES:
Complete response rate to navtemadlin, cytarabine and idarubicin | Up to 2 years
  Defined as (complete response [CR] without minimal residual disease [CR MRD negative(-ve)], CR or CR with incomplete hematologic recovery [CRi]). Will be based on the revised European LeukemiaNet (ELN) criteria (Dohner et al., 2017).
Complete cytogenetic response to navtemadlin, cytarabine and idarubicin | Up to 2 years
  Defined as cytogenic CR or molecular complete CR. Will be based on the revised ELN criteria (Dohner et al., 2017).
Progression-free survival (PFS) | From start of treatment to progression/recurrence or death - whichever comes first, assessed up to 2 years
  Patients who are alive and have not progressed or recurred at the time of their last disease assessment, will be censored at that time.
Pharmacodynamic (PD) effects of navtemadlin, in combination with induction chemotherapy on leukemia blasts | Up to 2 years
Potential predictive biomarkers of sensitivity to this regimen (MTF2/H3K27me3) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Kelly, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (6):
- United States (6):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT04190550/ICF_000.pdf